CLINICAL TRIAL: NCT01914939
Title: A Randomized, Controlled Trial of Intranasal Oxytocin as an Adjunct to Behavioral Therapy for Autism Spectrum Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Massachusetts Institute of Technology (Other)
Responsible Party: Principal Investigator, Aude Henin, Co-Director, Child CBT Program, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: W81XWH-12-1-0543; Clinical Trial Award (Other Grant/Funding Number: Department of Defense-Autism Research Program)
Record Dates: First submitted 2013-07-29; First posted 2013-08-02 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Autism Spectrum Disorders
Keywords: autism spectrum disorder; social skills deficits; cognitive behavioral therapy; oxytocin; young adult
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Oxytocin; Relaxation Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Social Skills Focused CBT (Experimental): Twelve weekly 60-minute sessions of social skills focused CBT
  Interventions: Behavioral: Social Skills focused CBT
- Stress Management/Relaxation Training (Active Comparator): Twelve weekly 60-minute sessions of stress management training
  Interventions: Behavioral: Stress management/relaxation training
- Oxytocin (Experimental): Intranasal administration of 24 IU of oxytocin
  Interventions: Drug: Oxytocin
- placebo drug (Placebo Comparator): Intranasal placebo drug
  Interventions: Drug: placebo drug

INTERVENTIONS:
Drug: Oxytocin
  Arms: Oxytocin
Behavioral: Social Skills focused CBT
  Arms: Social Skills Focused CBT
Behavioral: Stress management/relaxation training
  Arms: Stress Management/Relaxation Training
Drug: placebo drug
  Arms: placebo drug

SUMMARY:
This 3-year study is a trial of cognitive behavioral therapy (CBT), with or without oxytocin (OT) augmentation, in young adults with autism spectrum disorders. Participants will be randomly assigned to receive either a social skills-focused CBT intervention or a stress management/relaxation training CBT intervention. Participants will also be randomized to receive either a) intranasal oxytocin or b) a placebo drug, prior to the psychotherapy. The design of the study will enable examination of the efficacy of CBT for young adults with autism spectrum disorders. The design of the study will also allow examination of whether oxytocin enhances the efficacy of CBT.

The investigators will perform functional (fMRI) and structural (MRI) imaging with all participants prior to treatment. This will enable examination of the relations between measures of brain function and structure, and improvements in target symptoms over the course of treatment. The aim is to discover whether there are neural characteristics that can identify which participants with autism spectrum disorders are most likely to respond to CBT interventions and/or oxytocin treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40
* Able to attend in person therapy sessions in Boston
* Male
* English-speaking
* Normal or corrected vision
* No history of known genetic disorder, significant motor developmental difficulties, prematurity or brain injury
* IQ > 90, as determined by the WASI
* Score above the cutoff on the Reciprocal Social Interactions and the Restricted, Repetitive, and Stereotyped Behaviors Domains on the ADI-R, meet criteria for PDD or autism on the ADOS, and/or meet DSM-IV criteria for Autism Spectrum Disorder according to clinician interview.

Exclusion Criteria:

* Current use of certain endocrinologically relevant medications
* Current dependence on substances other than tobacco or caffeine
* History of serious medical illness, including neurological, endocrine, cardiac, respiratory, and metabolic diseases that are counter-indications to oxytocin
* Severe, current psychiatric disorder (ie, current mania, severe depression, psychosis, suicidality, severe aggression)
* Long QT, as determined by baseline EKG
* Current participation in other psychotherapy

Additional exclusion criteria for MRI scan only:

Participants who are MRI-ineligible will be enrolled in the clinical trial portion of the study, but will not undergo the MRI scan at MIT. Exclusion criteria for MRI are:

* Presence of metal implants or other metal in the body
* History of claustrophobia or inability to tolerate MRI

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2014-04; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Changes in the Autism Diagnostic Observation Schedule (ADOS) | At baseline and after 12 weeks of treatment
  The ADOS is a semi-structured standardized assessment of communication and social interaction that is considered a gold-standard assessment of autism spectrum disorders. The study will use Module 4, designed for use with adolescents and adults. The primary endpoint(dependent measure) will be the change in a global impression of social engagement by a clinician who is an experienced ADOS administrator. This will be a rating on a 10-point scale and involve expert clinical judgement of the qualities and behaviors that are at the core of the social/communicative deficits.
Clinical Global Impression Scale (CGI) | At baseline and every 4 week up to 12 weeks
  Independent Evaluator rated measure of autism symptom severity and improvement

SECONDARY OUTCOMES:
Social Responsiveness Scale (SRS) | At baseline and every 4 weeks up to 12 weeks
  65-item rating scale that measures the severity of autism spectrum symptoms
Reading the Mind in the Eyes Test (RMET) | At baseline and every 4 weeks up to 12 weeks
  Computerized measure of social skills
Social Ball Tossing Task | At baseline and every 4 weeks up to 12 weeks
  Computerized measure of social skills

OTHER OUTCOMES:
Self-Control Behavior Scale (SCBS) | At baseline and every 4 weeks up to 12 weeks
  Self-report questionnaire of coping and problem-solving skills
Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) | At baseline and every 4 weeks up to 12 weeks
  Self-report questionnaire of psychosocial functioning
Social Phobia and Anxiety Inventory (SPAI) | At baseline and every 4 weeks up to 12 weeks
  Self-report questionnaire of social anxiety
Social Adjustment Scale (SAS) | At baseline and every 4 weeks up to 12 weeks
  Self-report and parent-rated measure of psychosocial functioning
Vineland Adaptive Behavior Scales, 2nd Edition | At baseline and every 4 weeks up to 12 weeks
  Measure of adaptive and functional behaviors
Beck Depression Inventory (BDI) | At baseline and every 4 weeks up to 12 weeks
  Self-report questionnaire of depression symptoms
Global Assessment of Functioning (GAF) | At baseline and every 4 weeks up to 12 weeks
  Overall rating of impairment
Safety Monitoring Uniform Report Form | At baseline and every 4 weeks up to 12 weeks
  Assessment of adverse effects associated with oxytocin or placebo
Autism Diagnostic Interview-Revised (ADI-R) | Baseline
  Parent-report, clinician-administered assessment of autism spectrum disorder symptoms in their child
Structured Clinical Interview for DSM-IV (SCID) | Baseline
  A semistructured, clinician-administered assessment that assesses the presence of major psychiatric disorders. It is administered to the participant and to a parent about the participant.
Wechsler Intelligence Scales (WASI and WAIS-III) | Baseline
  Measures of current intellectual functioning. Will be used to assess inclusion/exclusion criteria.
Care Utilization | At baseline and every 4 weeks up to 12 weeks
  Assessment of any treatments (including medications, naturopathic treatments, speech or occupational therapy, hospitalizations, and intensive day programs) received over the past month.
Service Evaluation Questionnaire | After 12 weeks of treatment
  Self-report questionnaire about the participant's satisfaction with the psychosocial treatment they received.
Participant Adherence to the Intervention | after 12 weeks of treatment
  Information will be collected about a) the number of sessions attended by each participant; b) completion of homework assignments; and c) participation in the treatment sessions, using a 0-5 scale
Expectancy Rating Questionnaire | at week 1 of treatment
  Brief, self-report questionnaire about the participant's expectations of and belief in the social skills or stress management/relaxation interventions presented in the first session.
Adaptive Behavioral Assessment Scale-3rd edition | at weeks, 1, 4, 8, and 12
  self-report measure of adaptive functioning

CONTACTS AND LOCATIONS:
Overall Officials: John Gabrieli, PhD, Principal Investigator — Massachusetts General Hospital/MIT; Aude Henin, PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Massachusetts Institute of Technology Martinos Imaging Center, Cambridge, Massachusetts

REFERENCES:
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711